CLINICAL TRIAL: NCT00356226
Title: The Effects of Clonidine on the Diuretic Response in Cirrhotic Patients With Ascites and Activation of Sympathetic Nervous System: a Randomized Double-Blind Placebo Controlled Study.
Brief Title: The Effects of Clonidine on the Diuretic Response in Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Charleroi (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HEP-05-1550.R2
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2000-10

CONDITIONS: Ascitic Cirrhosis; Hyperactivation of Sympathetic Nervous System
Keywords: norepinephrine; renin; aldosterone; hemodynamics; spironolactone
MeSH Terms: interventions — Clonidine

INTERVENTIONS:
Drug: clonidine

SUMMARY:
To examine the effects of the addition of clonidine to diuretics on the mobilization of ascites at short-term (diuretic response and requirement of diuretics) and long-term (readmissions for tense ascites and requirement of diuretics) in cirrhotics with increased sympathetic nervous system. Secondary objectives were to study neuro-hormonal,hemodynamic effects and side effects of clonidine and diuretics.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with ascites
* Plasma norepinephrine level > 300 pg/mL (normal value: 185 - 275 pg/mL)

Exclusion Criteria:

* Serum bilirubin concentration above 4.5 mg/dL
* Prothrombin time below 40%
* Platelet count below 40 X 10¨9/liter
* Serum creatinine concentration above 2 mg/dL
* Gastro-intestinal hemorrhage
* Alcoholic hepatitis
* Diabetes mellitus,
* Hepatocellular carcinoma
* Respiratory or cardiac failures
* Hepatic encephalopathy
* Bacterial infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Lenaerts Anne, MD, Principal Investigator — ISPPC CHU de Charleroi
Locations (1):
- ISPPC CHU de Charleroi, Charleroi, Belgium

REFERENCES:
- [Background] Lenaerts A, Codden T, Henry JP, Legros F, Ligny G. Comparative pilot study of repeated large volume paracentesis vs the combination on clonidine-spironolactone in the treatment of cirrhosis-associated refractory ascites. Gastroenterol Clin Biol. 2005 Nov;29(11):1137-42. doi: 10.1016/s0399-8320(05)82178-5. PMID 16505759
- [Background] Lenaerts A, Codden T, Van Cauter J, Meunier JC, Henry JP, Ligny G. Interest of the association clonidine-spironolactone in cirrhotic patients with ascites and activation of sympathetic nervous system. Acta Gastroenterol Belg. 2002 Jan-Mar;65(1):1-5. PMID 12014310
- [Background] Lenaerts A, Codden T, Henry JP, Van Cauter J, Meunier JC, Ligny G. [Biological factors influencing response to diuretics in patients with cirrhosis and ascites]. Gastroenterol Clin Biol. 2001 Mar;25(3):268-72. French. PMID 11395674
- [Background] Lenaerts A, Van Cauter J, Moukaiber H, Meunier JC, Ligny G. [Treatment of refractory ascites with clonidine and spironolactone]. Gastroenterol Clin Biol. 1997;21(6-7):524-5. No abstract available. French. PMID 9295984
- [Result] Lenaerts A, Codden T, Meunier JC, Henry JP, Ligny G. Effects of clonidine on diuretic response in ascitic patients with cirrhosis and activation of sympathetic nervous system. Hepatology. 2006 Oct;44(4):844-9. doi: 10.1002/hep.21355. PMID 17006921